CLINICAL TRIAL: NCT05431114
Title: Quantitative MRI of Glenohumeral Cartilage & Labrum in Shoulder Instability
Acronym: OREF
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00110036
Record Dates: First submitted 2022-06-21; First posted 2022-06-24 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-04

CONDITIONS: Instability, Joint; Shoulder Dislocation; Shoulder Injuries; Shoulder Subluxation; Anterior Shoulder Instability; Glenoid; Dislocation
Keywords: Instability; Shoulder; Dislocation; Glenoid; Acute; Arthroscopy
MeSH Terms: conditions — Joint Instability; Shoulder Dislocation; Shoulder Injuries; Joint Dislocations

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Shoulder patients: Participants who presents with glenohumeral instability.
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Images of the injured shoulder will then be taken with magnetic resonance (MR) scanner. MRIs of each participant's shoulder will be acquired before and after completion of an exercise protocol.

SUMMARY:
The purpose of this study is to assess cartilage strain and contact areas following glenohumeral instability compared to healthy individuals.

DETAILED DESCRIPTION:
The purpose of this study is to assess cartilage strain and contact areas following glenohumeral instability compared to healthy individuals.

This is a prospective longitudinal cohort study to investigate cartilage strain and labral injury utilizing advance MRI techniques. Patients with shoulder instability will be studied at baseline (after injury and prior to surgical treatment) with glenohumeral cartilage strain MRI protocol, pre and post exercise. Patient reported outcomes including Western Ontario Shoulder Instability Index (WOSI), American Shoulder and Elbow Surgeon (ASES) Score, and PROMIS physical function and pain scores, will also be evaluated.

Data from this study will be compared to a previous study involving healthy controls that underwent the same exercises and imaging.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years old and ≤ 50 years old
* Acute injury involving anterior (front) shoulder dislocation
* Willingness to undergo arthroscopic shoulder stabilization
* Willingness to participant in standard rehabilitation

Exclusion Criteria:

* Moderate to severe osteoarthritis prior to surgery
* Will undergo bony augmentation to glenoid or humerus in addition to shoulder stabilization
* Unable to undergo standard pre and post-injury/operative rehabilitation
* History of inflammatory arthritis
* Previous surgery of the injured shoulder

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will consist of individuals ages 18 to 50 years old, who have sustained an anterior shoulder dislocation that requires surgical intervention.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Cartilage Strain at baseline | Baseline
  Cartilage strain will be assessed using images from MRIs.
Cartilage Strain at baseline at six months post-surgery | 6 months post-surgery
  Cartilage strain will be assessed using images from MRIs.
Western Ontario Shoulder Instability Index (WOSI) at baseline | Baseline
  The Western Ontario Shoulder Instability Index (WOSI) is an instability-specific patient reported outcome (PRO) measure for individuals with shoulder instability that was designed for use as a primary outcome measure in clinical trials evaluating treatments for patients with shoulder instability. The WOSI questionnaire consists of 21 items, each scored on a 100mm Visual Analogue Scale (VAS). Each item falls into one of the domains of physical function, sports/recreation/work, lifestyle and emotional well-being. Each question is scored between 0-100 points and the summation of all the questions results in a final WOSI score. The final score ranges from 0 (no decrease in shoulder-related quality of life) to 2100 (extreme distress in shoulder-related quality of life).
Western Ontario Shoulder Instability Index (WOSI) at six months post-surgery | 6 months post-surgery
  The Western Ontario Shoulder Instability Index (WOSI) is an instability-specific patient reported outcome (PRO) measure for individuals with shoulder instability that was designed for use as a primary outcome measure in clinical trials evaluating treatments for patients with shoulder instability. The WOSI questionnaire consists of 21 items, each scored on a 100mm Visual Analogue Scale (VAS). Each item falls into one of the domains of physical function, sports/recreation/work, lifestyle and emotional well-being. Each question is scored between 0-100 points and the summation of all the questions results in a final WOSI score. The final score ranges from 0 (no decrease in shoulder-related quality of life) to 2100 (extreme distress in shoulder-related quality of life).
American Shoulder and Elbow Surgeon (ASES) Score at baseline | Baseline
  The final American Shoulder and Elbow Surgeon (ASES) Score is obtained by summing the pain and functional portions with higher scores indicating better outcomes.
American Shoulder and Elbow Surgeon (ASES) Score at six months post-surgery | 6 months post-surgery
  The final American Shoulder and Elbow Surgeon (ASES) Score is obtained by summing the pain and functional portions with higher scores indicating better outcomes.
Patient-Reported Outcomes Measurement Information System (PROMIS) physical function at baseline | Baseline
  A PROMIS score of 50 is the average for the United States general population with a standard deviation of 10. A higher PROMIS T-score represents more of the concept being measured. For positively-worded concepts like Physical Function, Mobility, and Upper Extremity function, a T-score of 60 is one SD better than average. By comparison, a Physical Function T-score of 40 is one SD worse than average.
Patient-Reported Outcomes Measurement Information System (PROMIS) physical function at six months post-surgery | 6 months post-surgery
  A PROMIS score of 50 is the average for the United States general population with a standard deviation of 10. A higher PROMIS T-score represents more of the concept being measured. For positively-worded concepts like Physical Function, Mobility, and Upper Extremity function, a T-score of 60 is one SD better than average. By comparison, a Physical Function T-score of 40 is one SD worse than average.
Single Assessment Numeric Evaluation (SANE) Scores at baseline | Baseline
  The Single Assessment Numeric Evaluation (SANE) is a patient rating and is The SANE score represents one's perception of shoulder function as a percentage of normal, 0% being no function and 100% being normal function.
SANE Scores at six months post-surgery | 6 months post-surgery
  The Single Assessment Numeric Evaluation (SANE) is a patient rating and is The SANE score represents one's perception of shoulder function as a percentage of normal, 0% being no function and 100% being normal function.

SECONDARY OUTCOMES:
Correlation of labral injury and glenohumeral cartilage strain | Baseline & six months post-surgery
  The relationship between labral injury and glenohumeral cartilage strain and contact areas will be assessed using images from MRIs.
Change in cartilage strain and labrum following surgery | Six months post-surgery
  The relationship between labral injury and glenohumeral cartilage strain and contact areas will be assessed using images from MRIs from pre and post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Lau, MD, Principal Investigator — Duke University
Locations (1):
- Duke Sports Science Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No